CLINICAL TRIAL: NCT00959842
Title: Effects of Lovaza on Lipoprotein Composition and Function in Mild Hypertriglyceridemia
Acronym: ELLF
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanford Research (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, William S. Harris, Adjunct Senior Scientist, Sanford Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LVZ 112860; GSK - LVZ 112860 (Other Grant/Funding Number: GlaxoSmithKline)
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Results first posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-09

CONDITIONS: Hypertriglyceridemia
Keywords: hypertriglyceridemia; Omega-3 Fatty Acids; Lipoprotein; Statin; Lovaza
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Omacor; Fatty Acids, Omega-3; Fish Oils

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lovaza (Experimental): Lovaza was given as the only agent; there was no comparator agent or arm
  Interventions: Drug: Lovaza

INTERVENTIONS:
Drug: Lovaza — 1 gram gel capsule 4 capsules per day for 8 weeks
  Other Names: Omega-3 Fatty Acid; fish oil; Omacor

SUMMARY:
This study will build upon a previous finding that showed a triglyceride lowering effect of prescription omega-3 in combined therapy with statins. The proposed study will use a simple change from baseline design on 15 subjects who are hypertriglyceridemic on stable statin therapy. The protocol involves 3 study visits; each involve drawing a blood sample: day 1 - screening (blood draw for qualification and safety); day 7 - before taking prescription omega-3 fatty acids (Lovaza, 4 capsules/d; GlaxoSmithKline), day 63 -after taking prescription omega-3 fatty acids (Lovaza, 4 capsules/d; GlaxoSmithKline). The proposed study will include up to 15 subjects and will utilize several different measures of lipoprotein structure and function. The investigators will measure functional parameters such as the binding affinity of lipoproteins before and after treatment with omega-3 fatty acids. The investigators will also measure fatty acid, oxylipin and apolipoprotein content of plasma, very-low-density lipoprotein (VLDL), low-density lipoprotein (LDL) and high-density lipoprotein (HDL).

DETAILED DESCRIPTION:
This study will build upon a previous finding that showed a triglyceride lowering effect of prescription omega-3 in combined therapy with statins. The proposed study will use a simple change from baseline design on 15 subjects who are hypertriglyceridemic on stable statin therapy. The protocol involves 3 study visits; each involve drawing a blood sample: day 1 - screening (blood draw for qualification and safety); day 7 - before taking prescription omega-3 fatty acids (Lovaza, 4 capsules/d; GlaxoSmithKline), day 63 -after taking prescription omega-3 fatty acids (Lovaza, 4 capsules/d; GlaxoSmithKline). The proposed study will include up to 15 subjects and will utilize several different measures of lipoprotein structure and function. The investigators will measure functional parameters such as the binding affinity of lipoproteins before and after treatment with omega-3 fatty acids. The investigators will also measure fatty acid, oxylipin and apolipoprotein content of plasma, very-low-density lipoprotein (VLDL), low-density lipoprotein (LDL) and high-density lipoprotein (HDL).

ELIGIBILITY:
Inclusion Criteria:

* 18-79 years
* Stable does of statins ≥ 8 weeks prior to screening
* Good health by medical history, physical exam, electrocardiogram, laboratory test (e.g., serum chem., urinalysis)
* Mean fasting serum triglyceride of two most recent tests in medical record ≥ 200 and < 500 mg/dL
* Mean LDL-cholesterol of two most recent tests in medical record ≤ 1.1 × NCEP ATP III goal

Exclusion Criteria:

* Medications, vitamin pills, nutritional supplements or herbal preparations deemed exclusionary per primary investigator for possible interference
* Poorly controlled diabetes mellitus (e.g. [HbA1c] > 8.0%)
* History of a cardiovascular event
* Past revascularization procedure
* Past aortic aneurysm or an aortic dissection < 6 months prior to screening
* History of pancreatitis
* Sensitivity to any statin OR to omega-3 fatty acids or fish products
* Poorly controlled hypertension (i.e.: >=160 systolic (resting) and/or >=100 diastolic (resting)) at 2 consecutive visits
* Serum Creatinine ≥ 2.0 mg/dL
* Serum transaminase > 1.5 × upper limit of normal (ULN); including aspartate aminotransferase [AST] or alanine aminotransferase [ALT]; 31 U/L for AST, 45 U/L for ALT
* Creatine Kinase (CK) > 3.0 × ULN
* Taking other triglyceride lowering drugs (e.g., niacin, fibrates) or fish oil supplements providing more than 500 mg of EPA+DHA per day
* Contraindications for Lovaza per product insert
* Women who are pregnant or nursing

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory C Shearer, PhD, Principal Investigator — Sanford Research/USD
Locations (1):
- Sanford Research/USD, Sioux Falls, South Dakota, United States

REFERENCES:
- [Derived] Newman JW, Pedersen TL, Brandenburg VR, Harris WS, Shearer GC. Effect of omega-3 fatty acid ethyl esters on the oxylipin composition of lipoproteins in hypertriglyceridemic, statin-treated subjects. PLoS One. 2014 Nov 13;9(11):e111471. doi: 10.1371/journal.pone.0111471. eCollection 2014. PMID 25393536

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients on statins with persistent hypertriglyceridemia were identified by EMR search of hospital records. Letters were sent to eligible and those responding were screened and if qualifying, enrolled.
Pre-assignment Details: No run in or wash out
Period: Overall Study
Arm/Group | Lovaza
Started | 15 (17 were recruited and at baseline. 2 dropped out before starting the study drug. 15 finished)
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Lovaza: Lovaza was given as the only agent; there was no comparator agent or arm Lovaza: 1 gram gel capsule 4 capsules per day for 8 weeks
Arm/Group | Lovaza
Number analyzed (Participants) | 15
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 59 [46 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
lipids [Median (Inter-Quartile Range); unit: mg/dL]
  LDL-C | 88 [78 to 99]
  HDL-C | 38 [33 to 42]
  TG | 237 [200 to 270]

OUTCOME MEASURES:

1. Primary Outcome: HDL 15-HEPE
Description: high density lipoprotein level of 15-HEPE
Time Frame: 4 months
Population: hypertriglyceridemic statin treated patients
Measure: Mean (95% Confidence Interval); unit: nmol/mmol phospholipid
Arm/Group | Lovaza
Number analyzed (Participants) | 15
nmol/mmol phospholipid
  baseline | 3.7 [2.7 to 4.1]
  final | 10.4 [9.5 to 11]

ADVERSE EVENTS:
Groups:
- Treatment Group: all patients were treated with n3
Arm/Group | Treatment Group
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No